CLINICAL TRIAL: NCT01691859
Title: MEA115666: A Multi-centre, Open-label, Long Term Safety Study of Mepolizumab in Asthmatic Subjects Who Participated in the MEA112997 Trial
Brief Title: MEA112997 Open-label Long Term Extension Safety Study of Mepolizumab in Asthmatic Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115666; 2012-001643-51 (EudraCT Number)
Expanded Access: NCT00244686 (No longer available)
Record Dates: First submitted 2012-09-13; First posted 2012-09-25 (Estimated); Results first posted 2018-05-22 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Asthma
Keywords: extension study; Severe refractory asthma; safety; SB-240563; mepolizumab; eosinophils
MeSH Terms: conditions — Asthma | interventions — mepolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mepolizumab (Experimental): Subjects will receive 100 mg of mepolizumab (in 1ml polypropylene syringe) injected subcutaneously (SC) approximately every 4 weeks.
  Interventions: Drug: Mepolizumab

INTERVENTIONS:
Drug: Mepolizumab — 100 mg of mepolizumab will be injected subcutaneously (SC) once every 4 weeks

SUMMARY:
This is a multi-centre, open-label long term safety study of 100 milligrams (mg) mepolizumab administered subcutaneously (SC) in addition to standard of care in subjects who participated in the MEA112997 study. At each clinic visit, adverse events will be assessed and exacerbations will also be reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent.
* MEA112997 Study Participation: Received at least 2 doses of double-blind investigational product during the MEA112997 trial.
* MEA112997 Treatment Assignment: If the subject received mepolizumab, they must have had a positive risk: benefit ratio.
* Currently being treated with a controller medication and the subject has been on a controller medication for the past 12 weeks.
* Male or Eligible Female Subjects. To be eligible for entry into the study, females of childbearing potential must commit to consistent and correct use of an acceptable method of birth control for the duration of the trial and for 4 months after the last study drug administration.

Exclusion Criteria:

* Hypersensitivity related to mepolizumab.
* Clinically significant change in health status since completing participation in the MEA112997 trial.
* A current malignancy or previous history of cancer in remission for less than 12 months prior to screening.
* For those subjects who had a SAE in MEA112997 that was assessed as possibly related to mepolizumab by the investigator.
* Subjects who are pregnant or breastfeeding. Subjects should not be enrolled if they plan to become pregnant during the time of study participation.
* Screening ECG which has a clinically significant abnormality.
* Received Xolair (omalizumab) within the past 130 days.
* Participated in a clinical trial within the past 30 days or have received investigational medication within five terminal half-lives of Screen Visit, whichever is longer.
* Current smokers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2012-09-28 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (59):
- United States (11):
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Albany, Georgia
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
- Argentina (3):
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
- Australia (5):
  - GSK Investigational Site, New Lambton, New South Wales
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Canada (4):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Québec, Quebec
- Chile (4):
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Puente Alto - Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
  - GSK Investigational Site, Talcahuano
- France (4):
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Saint-Pierre
- Germany (6):
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Magdeburg
- Poland (2):
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Wroclaw
- Romania (3):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Târgu Mureş
- Russia (6):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, St'Petersburg
- South Korea (2):
  - GSK Investigational Site, Cheongju, Chungcheongbuk-do
  - GSK Investigational Site, Suwon, Kyonggi-do
- Ukraine (5):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
- United Kingdom (4):
  - GSK Investigational Site, Leicester, Leicestershire
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

REFERENCES:
- [Background] Khatri S, Moore W, Gibson PG, Leigh R, Bourdin A, Maspero J, Barros M, Buhl R, Howarth P, Albers FC, Bradford ES, Gilson M, Price RG, Yancey SW, Ortega H. Assessment of the long-term safety of mepolizumab and durability of clinical response in patients with severe eosinophilic asthma. J Allergy Clin Immunol. 2019 May;143(5):1742-1751.e7. doi: 10.1016/j.jaci.2018.09.033. Epub 2018 Oct 23. PMID 30359681
- [Derived] Ortega HG, Meyer E, Brusselle G, Asano K, Prazma CM, Albers FC, Mallett SA, Yancey SW, Gleich GJ. Update on immunogenicity in severe asthma: Experience with mepolizumab. J Allergy Clin Immunol Pract. 2019 Sep-Oct;7(7):2469-2475.e1. doi: 10.1016/j.jaip.2019.03.042. Epub 2019 Apr 5. No abstract available. PMID 30954640

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-center, open-label, long term safety study of mepolizumab in 347 asthmatic participants who participated in the MEA112997 trial and were found eligible for this study after screening and run in phase. The study was conducted at 65 centers in 13 countries from 28 Sep 2012 to 31 May 2017.
Pre-assignment Details: A total of 362 participants were screened; 4 participants were screen failures (did not meet the inclusion/exclusion criteria); 11 participants were withdrawn during the run-in period (4 did not meet the continuation criteria, 4 withdrawal by participant and 3 following physician decision).
Groups:
- Mepolizumab 100 mg: Participants received 100 milligram (mg) of mepolizumab injected subcutaneously (SC) once every 4 weeks until participant withdrawal or mepolizumab becomes commercially available in the relevant participating country. Participants remained on standard of care asthma therapy, which was adjusted during the study, at the discretion of their physician.
Period: Overall Study
Arm/Group | Mepolizumab 100 mg
Started | 347
Completed | 0
Not Completed | 347
Not completed — Adverse Event | 19
Not completed — Lack of Efficacy | 11
Not completed — Protocol Violation | 4
Not completed — Product commercially available | 221
Not completed — Study closed/terminated | 50
Not completed — Lost to Follow-up | 5
Not completed — Physician Decision | 6
Not completed — Withdrawal by Subject | 31

BASELINE CHARACTERISTICS:
Groups:
- Mepolizumab 100 mg: Participants received 100 mg of mepolizumab injected SC once every 4 weeks until participant withdrawal or mepolizumab becomes commercially available in the relevant participating country. Participants remained on standard of care asthma therapy, which was adjusted during the study, at the discretion of their physician.
Arm/Group | Mepolizumab 100 mg
Number analyzed (Participants) | 347
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.2 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 224
  Male | 123
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 8
  American Indian or Alaskan Native | 2
  Asian - Central/South Asian Heritage | 4
  Asian - East Asian Heritage | 14
  White - Arabic/North African Heritage | 7
  White - White/Caucasian/European Heritage | 311
  Asian & Native Hawaiian or Other Pacific Islander | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced On-treatment Adverse Events (AE) and On-treatment Serious Adverse Events (SAE)
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with use of a medicinal product (MP), whether or not considered related to MP. AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with use of MP. SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant or all events of possible drug induced liver injury with hyperbilirubinemia. As Treated (AT) Population consisted of participants who received at least one dose of open label mepolizumab. On-treatment AEs and on-treatment SAEs are the events occurring on/after the first dose of open-label mepolizumab date and before/on last dose of mepolizumab + 28 days.
Time Frame: Baseline (Week 0) to Week 240
Population: AT Population.
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 100 mg
Number analyzed (Participants) | 347
Participants
  AE | 326
  SAE | 79

2. Secondary Outcome: Number of Participants Who Experienced On-treatment Systemic (i.e., Allergic/Immunoglobulin E [IgE]-Mediated and Non-allergic) and On-treatment Local Site Reactions
Description: Systemic and local site reactions following mepolizumab dosing as identified by the investigator and the number of participants who experienced systemic and/or local site reactions are presented. On-treatment AEs and on-treatment SAEs are the events occurring on/after the first dose of open-label mepolizumab date and before/on last dose of mepolizumab + 28 days.
Time Frame: Baseline (Week 0) to Week 240
Population: AT Population.
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 100 mg
Number analyzed (Participants) | 347
Participants
  Systemic reactions | 9
  Local site reactions | 42

3. Secondary Outcome: Mean Change From Baseline in QT Interval Corrected by Bazett's Method (QTc[B])
Description: Twelve-lead ECGs were performed at Screening and every 24 weeks during the treatment period. ECG measurements were made after the participant had rested in the supine position for 5 minutes. Collection shortly after a meal or during sleep was avoided as QT prolongation can occur at these times. Baseline was the last available ECG prior to mepolizumab dosing. Change from Baseline was post-Baseline values minus Baseline values. Only those participants available at the specified time points were analyzed represented by n=X in the category titles.
Time Frame: Baseline (Week 0) to Week 240
Population: AT Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Mepolizumab 100 mg
Number analyzed (Participants) | 347
Milliseconds
  Week 24, n=330: number analyzed (Participants) | 330
  Week 24, n=330 | 4.2 (18.57)
  Week 48, n=319: number analyzed (Participants) | 319
  Week 48, n=319 | 3.2 (17.19)
  Week 72, n=307: number analyzed (Participants) | 307
  Week 72, n=307 | -0.5 (16.76)
  Week 96, n=293: number analyzed (Participants) | 293
  Week 96, n=293 | 1.3 (17.92)
  Week 124, n=292: number analyzed (Participants) | 292
  Week 124, n=292 | 1.5 (19.69)
  Week 148, n=275: number analyzed (Participants) | 275
  Week 148, n=275 | 1.6 (17.84)
  Week 176, n=201: number analyzed (Participants) | 201
  Week 176, n=201 | 0.6 (18.02)
  Week 200, n=149: number analyzed (Participants) | 149
  Week 200, n=149 | 3.3 (17.02)
  Week 228, n=32: number analyzed (Participants) | 32
  Week 228, n=32 | 1.5 (20.95)
  Follow up, n=270: number analyzed (Participants) | 270
  Follow up, n=270 | 2.5 (18.71)

4. Secondary Outcome: Mean Change From Baseline in QT Interval Corrected by Fridericia's Method (QTc[F])
Description: as for outcome 3
Time Frame: Baseline (Week 0) to Week 240
Population: AT Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Mepolizumab 100 mg
Number analyzed (Participants) | 347
Milliseconds
  Week 24, n=330: number analyzed (Participants) | 330
  Week 24, n=330 | 5.1 (17.00)
  Week 48, n=319: number analyzed (Participants) | 319
  Week 48, n=319 | 4.1 (15.72)
  Week 72, n=307: number analyzed (Participants) | 307
  Week 72, n=307 | 0.2 (15.11)
  Week 96, n=293: number analyzed (Participants) | 293
  Week 96, n=293 | 2.2 (15.37)
  Week 124, n=292: number analyzed (Participants) | 292
  Week 124, n=292 | 3.2 (16.77)
  Week 148, n=275: number analyzed (Participants) | 275
  Week 148, n=275 | 2.9 (15.49)
  Week 176, n=201: number analyzed (Participants) | 201
  Week 176, n=201 | 2.0 (15.97)
  Week 200, n=149: number analyzed (Participants) | 149
  Week 200, n=149 | 4.3 (14.52)
  Week 228, n=32: number analyzed (Participants) | 32
  Week 228, n=32 | 0.4 (15.81)
  Follow up, n=270: number analyzed (Participants) | 270
  Follow up, n=270 | 3.9 (16.39)

5. Secondary Outcome: Number of Participants With a Maximum Change From Baseline for QTc(F) and QTc(B)
Description: Twelve-lead ECGs were performed at Screening and every 24 weeks during the treatment period. ECG measurements were made after the participant had rested in the supine position for 5 minutes. Collection shortly after a meal or during sleep was avoided as QT prolongation can occur at these times. Baseline was the last available ECG prior to mepolizumab dosing. Change from Baseline was post-Baseline values minus Baseline values. Number of participants with a maximum change from Baseline for QTc(F) and QTc(B) at any time post Baseline are presented. Only those participants who provided ECG data at baseline and post-baseline were analyzed.
Time Frame: Baseline (Week 0) to Week 240
Population: AT Population.
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 100 mg
Number analyzed (Participants) | 342
Participants
  QTc(F): < -60 | 0
  QTc(F): >= -60 - < -30 | 1
  QTc(F): >= -30 - < 0 | 31
  QTc(F): >= 0 - < 30 | 252
  QTc(F): >= 30 - < 60 | 55
  QTc(F): >= 60 | 3
  QTc(B): < -60 | 0
  QTc(B): >= -60 - < -30 | 1
  QTc(B): >= -30 - < 0 | 36
  QTc(B): >= 0 - < 30 | 228
  QTc(B): >= 30 - < 60 | 69
  QTc(B): >= 60 | 8

6. Secondary Outcome: Number of Participants With Clinical Chemistry Data of Potential Clinical Concern
Description: Clinical chemistry analytes with laboratory ranges defining values of potential clinical concern included sodium, potassium, calcium, phosphate, serum glucose and alanine aminotransferase. Number of participants with clinical chemistry abnormalities of potential clinical concern anytime post baseline are presented. Only those participants who provided lab data post-baseline were analyzed represented by n=X in the category titles.
Time Frame: Baseline (Week 0) to Week 240
Population: AT Population.
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 100 mg
Number analyzed (Participants) | 346
Participants
  Potassium high, n=346 | 1
  Serum glucose high, n=346 | 1
  Serum glucose low, n=346 | 7

7. Secondary Outcome: Number of Participants With Hematology Data of Potential Clinical Concern
Description: Hematology parameters with laboratory ranges defining values of potential clinical concern included hemoglobin, hematocrit, platelet count, white blood cell count. Number of participants with clinical hematology abnormalities of potential clinical concern anytime post baseline are presented, which only included participants with low hemoglobin values. Only those participants who provided lab data post-baseline were analyzed.
Time Frame: Baseline (Week 0) to Week 240
Population: AT Population.
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 100 mg
Number analyzed (Participants) | 346
Participants | 1

8. Secondary Outcome: Mean Change From Baseline in Vital Signs-Sitting Diastolic Blood Pressure and Sitting Systolic Blood Pressure
Description: Vital signs included sitting pulse rate and sitting blood pressure (diastolic and systolic). Measurements were done pre injection with the participant sitting, having rested in this position for at least 5 minutes before each reading. Baseline was Week 0. Change from Baseline was post-Baseline values minus Baseline values. Only those participants available at the specified time points were analyzed represented by n=X in the category titles.
Time Frame: Baseline (Week 0) to Week 240
Population: AT Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Mepolizumab 100 mg
Number analyzed (Participants) | 347
Millimeters of mercury (mmHg)
  Sitting Diastolic Blood Pressure: Week 4, n=346: number analyzed (Participants) | 346
  Sitting Diastolic Blood Pressure: Week 4, n=346 | -1.0 (8.71)
  Sitting Diastolic Blood Pressure: Week 8, n=345: number analyzed (Participants) | 345
  Sitting Diastolic Blood Pressure: Week 8, n=345 | -1.5 (8.85)
  Sitting Diastolic Blood Pressure: Week 12, n=342: number analyzed (Participants) | 342
  Sitting Diastolic Blood Pressure: Week 12, n=342 | -0.7 (9.67)
  Sitting Diastolic Blood Pressure: Week 16, n=341: number analyzed (Participants) | 341
  Sitting Diastolic Blood Pressure: Week 16, n=341 | -1.6 (9.27)
  Sitting Diastolic Blood Pressure: Week 20, n=338: number analyzed (Participants) | 338
  Sitting Diastolic Blood Pressure: Week 20, n=338 | -1.6 (9.17)
  Sitting Diastolic Blood Pressure: Week 24, n=336: number analyzed (Participants) | 336
  Sitting Diastolic Blood Pressure: Week 24, n=336 | -0.7 (9.27)
  Sitting Diastolic Blood Pressure: Week 28, n=332: number analyzed (Participants) | 332
  Sitting Diastolic Blood Pressure: Week 28, n=332 | -1.3 (8.90)
  Sitting Diastolic Blood Pressure: Week 32, n=333: number analyzed (Participants) | 333
  Sitting Diastolic Blood Pressure: Week 32, n=333 | -1.0 (9.62)
  Sitting Diastolic Blood Pressure: Week 36, n=329: number analyzed (Participants) | 329
  Sitting Diastolic Blood Pressure: Week 36, n=329 | -1.8 (8.95)
  Sitting Diastolic Blood Pressure: Week 40, n=329: number analyzed (Participants) | 329
  Sitting Diastolic Blood Pressure: Week 40, n=329 | -1.2 (9.33)
  Sitting Diastolic Blood Pressure: Week 44, n=326: number analyzed (Participants) | 326
  Sitting Diastolic Blood Pressure: Week 44, n=326 | -1.1 (10.00)
  Sitting Diastolic Blood Pressure: Week 48, n=325: number analyzed (Participants) | 325
  Sitting Diastolic Blood Pressure: Week 48, n=325 | -0.7 (9.67)
  Sitting Diastolic Blood Pressure: Week 52, n=322: number analyzed (Participants) | 322
  Sitting Diastolic Blood Pressure: Week 52, n=322 | -1.1 (9.85)
  Sitting Diastolic Blood Pressure: Week 56, n=320: number analyzed (Participants) | 320
  Sitting Diastolic Blood Pressure: Week 56, n=320 | -1.3 (9.67)
  Sitting Diastolic Blood Pressure: Week 60, n=318: number analyzed (Participants) | 318
  Sitting Diastolic Blood Pressure: Week 60, n=318 | -0.9 (9.56)
  Sitting Diastolic Blood Pressure: Week 64, n=318: number analyzed (Participants) | 318
  Sitting Diastolic Blood Pressure: Week 64, n=318 | -1.0 (9.29)
  Sitting Diastolic Blood Pressure: Week 68, n=317: number analyzed (Participants) | 317
  Sitting Diastolic Blood Pressure: Week 68, n=317 | -1.1 (9.94)
  Sitting Diastolic Blood Pressure: Week 72, n=312: number analyzed (Participants) | 312
  Sitting Diastolic Blood Pressure: Week 72, n=312 | -1.5 (9.67)
  Sitting Diastolic Blood Pressure: Week 76, n=313: number analyzed (Participants) | 313
  Sitting Diastolic Blood Pressure: Week 76, n=313 | -1.1 (10.06)
  Sitting Diastolic Blood Pressure: Week 80, n=311: number analyzed (Participants) | 311
  Sitting Diastolic Blood Pressure: Week 80, n=311 | -1.6 (10.23)
  Sitting Diastolic Blood Pressure: Week 84, n=310: number analyzed (Participants) | 310
  Sitting Diastolic Blood Pressure: Week 84, n=310 | -1.7 (10.51)
  Sitting Diastolic Blood Pressure: Week 88, n=310: number analyzed (Participants) | 310
  Sitting Diastolic Blood Pressure: Week 88, n=310 | -1.4 (10.45)
  Sitting Diastolic Blood Pressure: Week 92, n=311: number analyzed (Participants) | 311
  Sitting Diastolic Blood Pressure: Week 92, n=311 | -1.0 (9.89)
  Sitting Diastolic Blood Pressure: Week 96, n=303: number analyzed (Participants) | 303
  Sitting Diastolic Blood Pressure: Week 96, n=303 | -1.2 (9.81)
  Sitting Diastolic Blood Pressure: Week 100, n=300: number analyzed (Participants) | 300
  Sitting Diastolic Blood Pressure: Week 100, n=300 | -0.3 (9.40)
  Sitting Diastolic Blood Pressure: Week 104, n=301: number analyzed (Participants) | 301
  Sitting Diastolic Blood Pressure: Week 104, n=301 | -1.0 (9.69)
  Sitting Diastolic Blood Pressure: Week 108, n=300: number analyzed (Participants) | 300
  Sitting Diastolic Blood Pressure: Week 108, n=300 | -0.9 (10.28)
  Sitting Diastolic Blood Pressure: Week 112, n=299: number analyzed (Participants) | 299
  Sitting Diastolic Blood Pressure: Week 112, n=299 | -0.9 (9.78)
  Sitting Diastolic Blood Pressure: Week 116, n=297: number analyzed (Participants) | 297
  Sitting Diastolic Blood Pressure: Week 116, n=297 | -0.7 (9.56)
  Sitting Diastolic Blood Pressure: Week 120, n=295: number analyzed (Participants) | 295
  Sitting Diastolic Blood Pressure: Week 120, n=295 | -0.8 (9.41)
  Sitting Diastolic Blood Pressure: Week 124, n=294: number analyzed (Participants) | 294
  Sitting Diastolic Blood Pressure: Week 124, n=294 | -1.3 (10.52)
  Sitting Diastolic Blood Pressure: Week 128, n=293: number analyzed (Participants) | 293
  Sitting Diastolic Blood Pressure: Week 128, n=293 | -1.2 (10.08)
  Sitting Diastolic Blood Pressure: Week 132, n=289: number analyzed (Participants) | 289
  Sitting Diastolic Blood Pressure: Week 132, n=289 | -1.0 (10.48)
  Sitting Diastolic Blood Pressure: Week 136, n=288: number analyzed (Participants) | 288
  Sitting Diastolic Blood Pressure: Week 136, n=288 | -0.7 (10.42)
  Sitting Diastolic Blood Pressure: Week 140, n=287: number analyzed (Participants) | 287
  Sitting Diastolic Blood Pressure: Week 140, n=287 | -0.6 (9.90)
  Sitting Diastolic Blood Pressure: Week 144, n=290: number analyzed (Participants) | 290
  Sitting Diastolic Blood Pressure: Week 144, n=290 | -0.9 (9.83)
  Sitting Diastolic Blood Pressure: Week 148, n=287: number analyzed (Participants) | 287
  Sitting Diastolic Blood Pressure: Week 148, n=287 | 0.1 (10.22)
  Sitting Diastolic Blood Pressure: Week 152, n=284: number analyzed (Participants) | 284
  Sitting Diastolic Blood Pressure: Week 152, n=284 | -0.9 (10.17)
  Sitting Diastolic Blood Pressure: Week 156, n=275: number analyzed (Participants) | 275
  Sitting Diastolic Blood Pressure: Week 156, n=275 | -0.4 (10.44)
  Sitting Diastolic Blood Pressure: Week 160, n=265: number analyzed (Participants) | 265
  Sitting Diastolic Blood Pressure: Week 160, n=265 | -0.6 (9.93)
  Sitting Diastolic Blood Pressure: Week 164, n=242: number analyzed (Participants) | 242
  Sitting Diastolic Blood Pressure: Week 164, n=242 | -1.7 (10.83)
  Sitting Diastolic Blood Pressure: Week 168, n=232: number analyzed (Participants) | 232
  Sitting Diastolic Blood Pressure: Week 168, n=232 | -1.3 (10.46)
  Sitting Diastolic Blood Pressure: Week 172, n=226: number analyzed (Participants) | 226
  Sitting Diastolic Blood Pressure: Week 172, n=226 | -1.2 (10.18)
  Sitting Diastolic Blood Pressure: Week 176, n=212: number analyzed (Participants) | 212
  Sitting Diastolic Blood Pressure: Week 176, n=212 | -1.6 (9.84)
  Sitting Diastolic Blood Pressure: Week 180, n=200: number analyzed (Participants) | 200
  Sitting Diastolic Blood Pressure: Week 180, n=200 | -1.6 (10.42)
  Sitting Diastolic Blood Pressure: Week 184, n=184: number analyzed (Participants) | 184
  Sitting Diastolic Blood Pressure: Week 184, n=184 | -1.3 (9.94)
  Sitting Diastolic Blood Pressure: Week 188, n=180: number analyzed (Participants) | 180
  Sitting Diastolic Blood Pressure: Week 188, n=180 | -1.4 (9.81)
  Sitting Diastolic Blood Pressure: Week 192, n=176: number analyzed (Participants) | 176
  Sitting Diastolic Blood Pressure: Week 192, n=176 | -1.1 (10.25)
  Sitting Diastolic Blood Pressure: Week 196, n=175: number analyzed (Participants) | 175
  Sitting Diastolic Blood Pressure: Week 196, n=175 | -1.5 (10.18)
  Sitting Diastolic Blood Pressure: Week 200, n=172: number analyzed (Participants) | 172
  Sitting Diastolic Blood Pressure: Week 200, n=172 | -0.4 (10.07)
  Sitting Diastolic Blood Pressure: Week 204, n=169: number analyzed (Participants) | 169
  Sitting Diastolic Blood Pressure: Week 204, n=169 | -1.1 (10.25)
  Sitting Diastolic Blood Pressure: Week 208, n=157: number analyzed (Participants) | 157
  Sitting Diastolic Blood Pressure: Week 208, n=157 | -1.8 (9.48)
  Sitting Diastolic Blood Pressure: Week 212, n=146: number analyzed (Participants) | 146
  Sitting Diastolic Blood Pressure: Week 212, n=146 | -1.3 (9.53)
  Sitting Diastolic Blood Pressure: Week 216, n=130: number analyzed (Participants) | 130
  Sitting Diastolic Blood Pressure: Week 216, n=130 | -0.2 (9.55)
  Sitting Diastolic Blood Pressure: Week 220, n=67: number analyzed (Participants) | 67
  Sitting Diastolic Blood Pressure: Week 220, n=67 | -1.6 (10.85)
  Sitting Diastolic Blood Pressure: Week 224, n=54: number analyzed (Participants) | 54
  Sitting Diastolic Blood Pressure: Week 224, n=54 | -1.9 (11.97)
  Sitting Diastolic Blood Pressure: Week 228, n=37: number analyzed (Participants) | 37
  Sitting Diastolic Blood Pressure: Week 228, n=37 | -0.2 (9.60)
  Sitting Diastolic Blood Pressure: Week 232, n=5: number analyzed (Participants) | 5
  Sitting Diastolic Blood Pressure: Week 232, n=5 | 4.6 (5.86)
  Sitting Diastolic Blood Pressure: Follow-up, n=306: number analyzed (Participants) | 306
  Sitting Diastolic Blood Pressure: Follow-up, n=306 | -0.7 (10.03)
  Sitting Systolic Blood Pressure: Week 4, n=346: number analyzed (Participants) | 346
  Sitting Systolic Blood Pressure: Week 4, n=346 | 0.2 (10.79)
  Sitting Systolic Blood Pressure: Week 8, n=345: number analyzed (Participants) | 345
  Sitting Systolic Blood Pressure: Week 8, n=345 | -0.7 (12.57)
  Sitting Systolic Blood Pressure: Week 12, n=342: number analyzed (Participants) | 342
  Sitting Systolic Blood Pressure: Week 12, n=342 | -0.3 (12.59)
  Sitting Systolic Blood Pressure: Week 16, n=341: number analyzed (Participants) | 341
  Sitting Systolic Blood Pressure: Week 16, n=341 | -0.5 (13.60)
  Sitting Systolic Blood Pressure: Week 20, n=338: number analyzed (Participants) | 338
  Sitting Systolic Blood Pressure: Week 20, n=338 | -1.8 (13.31)
  Sitting Systolic Blood Pressure: Week 24, n=336: number analyzed (Participants) | 336
  Sitting Systolic Blood Pressure: Week 24, n=336 | -0.8 (13.93)
  Sitting Systolic Blood Pressure: Week 28, n=332: number analyzed (Participants) | 332
  Sitting Systolic Blood Pressure: Week 28, n=332 | -0.6 (13.61)
  Sitting Systolic Blood Pressure: Week 32, n=333: number analyzed (Participants) | 333
  Sitting Systolic Blood Pressure: Week 32, n=333 | -1.0 (14.24)
  Sitting Systolic Blood Pressure: Week 36, n=329: number analyzed (Participants) | 329
  Sitting Systolic Blood Pressure: Week 36, n=329 | -0.7 (14.19)
  Sitting Systolic Blood Pressure: Week 40, n=329: number analyzed (Participants) | 329
  Sitting Systolic Blood Pressure: Week 40, n=329 | -0.6 (14.11)
  Sitting Systolic Blood Pressure: Week 44, n=326: number analyzed (Participants) | 326
  Sitting Systolic Blood Pressure: Week 44, n=326 | -0.9 (14.87)
  Sitting Systolic Blood Pressure: Week 48, n=325: number analyzed (Participants) | 325
  Sitting Systolic Blood Pressure: Week 48, n=325 | -0.1 (13.59)
  Sitting Systolic Blood Pressure: Week 52, n=322: number analyzed (Participants) | 322
  Sitting Systolic Blood Pressure: Week 52, n=322 | -0.3 (13.63)
  Sitting Systolic Blood Pressure: Week 56, n=320: number analyzed (Participants) | 320
  Sitting Systolic Blood Pressure: Week 56, n=320 | -0.3 (14.33)
  Sitting Systolic Blood Pressure: Week 60, n=318: number analyzed (Participants) | 318
  Sitting Systolic Blood Pressure: Week 60, n=318 | -0.0 (14.21)
  Sitting Systolic Blood Pressure: Week 64, n=318: number analyzed (Participants) | 318
  Sitting Systolic Blood Pressure: Week 64, n=318 | -0.2 (13.99)
  Sitting Systolic Blood Pressure: Week 68, n=317: number analyzed (Participants) | 317
  Sitting Systolic Blood Pressure: Week 68, n=317 | -1.1 (14.83)
  Sitting Systolic Blood Pressure: Week 72, n=312: number analyzed (Participants) | 312
  Sitting Systolic Blood Pressure: Week 72, n=312 | -1.8 (13.16)
  Sitting Systolic Blood Pressure: Week 76, n=313: number analyzed (Participants) | 313
  Sitting Systolic Blood Pressure: Week 76, n=313 | -0.8 (14.44)
  Sitting Systolic Blood Pressure: Week 80, n=311: number analyzed (Participants) | 311
  Sitting Systolic Blood Pressure: Week 80, n=311 | -1.1 (14.49)
  Sitting Systolic Blood Pressure: Week 84, n=310: number analyzed (Participants) | 310
  Sitting Systolic Blood Pressure: Week 84, n=310 | -1.9 (14.47)
  Sitting Systolic Blood Pressure: Week 88, n=310: number analyzed (Participants) | 310
  Sitting Systolic Blood Pressure: Week 88, n=310 | -1.7 (14.94)
  Sitting Systolic Blood Pressure: Week 92, n=311: number analyzed (Participants) | 311
  Sitting Systolic Blood Pressure: Week 92, n=311 | -0.3 (15.16)
  Sitting Systolic Blood Pressure: Week 96, n=303: number analyzed (Participants) | 303
  Sitting Systolic Blood Pressure: Week 96, n=303 | 0.1 (14.32)
  Sitting Systolic Blood Pressure: Week 100, n=300: number analyzed (Participants) | 300
  Sitting Systolic Blood Pressure: Week 100, n=300 | 0.7 (14.71)
  Sitting Systolic Blood Pressure: Week 104, n=301: number analyzed (Participants) | 301
  Sitting Systolic Blood Pressure: Week 104, n=301 | 0.3 (14.81)
  Sitting Systolic Blood Pressure: Week 108, n=300: number analyzed (Participants) | 300
  Sitting Systolic Blood Pressure: Week 108, n=300 | 0.5 (15.15)
  Sitting Systolic Blood Pressure: Week 112, n=299: number analyzed (Participants) | 299
  Sitting Systolic Blood Pressure: Week 112, n=299 | -0.4 (14.83)
  Sitting Systolic Blood Pressure: Week 116, n=297: number analyzed (Participants) | 297
  Sitting Systolic Blood Pressure: Week 116, n=297 | 0.4 (14.31)
  Sitting Systolic Blood Pressure: Week 120, n=295: number analyzed (Participants) | 295
  Sitting Systolic Blood Pressure: Week 120, n=295 | 0.5 (14.37)
  Sitting Systolic Blood Pressure: Week 124, n=294: number analyzed (Participants) | 294
  Sitting Systolic Blood Pressure: Week 124, n=294 | 0.7 (14.80)
  Sitting Systolic Blood Pressure: Week 128, n=293: number analyzed (Participants) | 293
  Sitting Systolic Blood Pressure: Week 128, n=293 | 0.7 (14.68)
  Sitting Systolic Blood Pressure: Week 132, n=289: number analyzed (Participants) | 289
  Sitting Systolic Blood Pressure: Week 132, n=289 | 0.7 (14.51)
  Sitting Systolic Blood Pressure: Week 136, n=288: number analyzed (Participants) | 288
  Sitting Systolic Blood Pressure: Week 136, n=288 | 0.9 (16.81)
  Sitting Systolic Blood Pressure: Week 140, n=287: number analyzed (Participants) | 287
  Sitting Systolic Blood Pressure: Week 140, n=287 | 0.3 (15.48)
  Sitting Systolic Blood Pressure: Week 144, n=290: number analyzed (Participants) | 290
  Sitting Systolic Blood Pressure: Week 144, n=290 | 1.1 (15.79)
  Sitting Systolic Blood Pressure: Week 148, n=287: number analyzed (Participants) | 287
  Sitting Systolic Blood Pressure: Week 148, n=287 | 1.8 (13.59)
  Sitting Systolic Blood Pressure: Week 152, n=284: number analyzed (Participants) | 284
  Sitting Systolic Blood Pressure: Week 152, n=284 | 0.2 (15.53)
  Sitting Systolic Blood Pressure: Week 156, n=275: number analyzed (Participants) | 275
  Sitting Systolic Blood Pressure: Week 156, n=275 | 0.8 (14.56)
  Sitting Systolic Blood Pressure: Week 160, n=265: number analyzed (Participants) | 265
  Sitting Systolic Blood Pressure: Week 160, n=265 | 1.1 (15.34)
  Sitting Systolic Blood Pressure: Week 164, n=242: number analyzed (Participants) | 242
  Sitting Systolic Blood Pressure: Week 164, n=242 | 0.6 (15.51)
  Sitting Systolic Blood Pressure: Week 168, n=232: number analyzed (Participants) | 232
  Sitting Systolic Blood Pressure: Week 168, n=232 | 0.1 (14.87)
  Sitting Systolic Blood Pressure: Week 172, n=226: number analyzed (Participants) | 226
  Sitting Systolic Blood Pressure: Week 172, n=226 | -0.8 (15.67)
  Sitting Systolic Blood Pressure: Week 176, n=212: number analyzed (Participants) | 212
  Sitting Systolic Blood Pressure: Week 176, n=212 | 0.4 (13.78)
  Sitting Systolic Blood Pressure: Week 180, n=200: number analyzed (Participants) | 200
  Sitting Systolic Blood Pressure: Week 180, n=200 | 0.6 (15.32)
  Sitting Systolic Blood Pressure: Week 184, n=184: number analyzed (Participants) | 184
  Sitting Systolic Blood Pressure: Week 184, n=184 | -0.5 (16.36)
  Sitting Systolic Blood Pressure: Week 188, n=180: number analyzed (Participants) | 180
  Sitting Systolic Blood Pressure: Week 188, n=180 | -1.0 (15.54)
  Sitting Systolic Blood Pressure: Week 192, n=176: number analyzed (Participants) | 176
  Sitting Systolic Blood Pressure: Week 192, n=176 | -1.2 (16.60)
  Sitting Systolic Blood Pressure: Week 196, n=175: number analyzed (Participants) | 175
  Sitting Systolic Blood Pressure: Week 196, n=175 | -0.8 (14.76)
  Sitting Systolic Blood Pressure: Week 200, n=172: number analyzed (Participants) | 172
  Sitting Systolic Blood Pressure: Week 200, n=172 | -0.1 (15.28)
  Sitting Systolic Blood Pressure: Week 204, n=169: number analyzed (Participants) | 169
  Sitting Systolic Blood Pressure: Week 204, n=169 | -0.4 (15.64)
  Sitting Systolic Blood Pressure: Week 208, n=157: number analyzed (Participants) | 157
  Sitting Systolic Blood Pressure: Week 208, n=157 | -1.0 (16.92)
  Sitting Systolic Blood Pressure: Week 212, n=146: number analyzed (Participants) | 146
  Sitting Systolic Blood Pressure: Week 212, n=146 | 0.5 (14.98)
  Sitting Systolic Blood Pressure: Week 216, n=130: number analyzed (Participants) | 130
  Sitting Systolic Blood Pressure: Week 216, n=130 | 0.4 (15.52)
  Sitting Systolic Blood Pressure: Week 220, n=67: number analyzed (Participants) | 67
  Sitting Systolic Blood Pressure: Week 220, n=67 | -4.2 (20.86)
  Sitting Systolic Blood Pressure: Week 224, n=54: number analyzed (Participants) | 54
  Sitting Systolic Blood Pressure: Week 224, n=54 | -3.8 (17.87)
  Sitting Systolic Blood Pressure: Week 228, n=37: number analyzed (Participants) | 37
  Sitting Systolic Blood Pressure: Week 228, n=37 | -3.6 (15.15)
  Sitting Systolic Blood Pressure: Week 232, n=5: number analyzed (Participants) | 5
  Sitting Systolic Blood Pressure: Week 232, n=5 | -0.8 (6.30)
  Sitting Systolic Blood Pressure: Follow-up, n=306: number analyzed (Participants) | 306
  Sitting Systolic Blood Pressure: Follow-up, n=306 | -0.0 (14.92)

9. Secondary Outcome: Mean Change From Baseline in Vital Signs-Sitting Pulse Rate
Description: Vital signs included sitting pulse rate and blood pressure (diastolic and systolic). Measurements were done pre injection with the participant sitting, having rested in this position for at least 5 minutes before each reading. Baseline was Week 0. Change from Baseline was post-Baseline values minus Baseline values. Only those participants available at the specified time points were analyzed represented by n=X in the category titles.
Time Frame: Baseline (Week 0) to Week 240
Population: AT Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Mepolizumab 100 mg
Number analyzed (Participants) | 347
Beats per minute
  Sitting Pulse Rate: Week 4, n=346: number analyzed (Participants) | 346
  Sitting Pulse Rate: Week 4, n=346 | -0.3 (8.94)
  Sitting Pulse Rate: Week 8, n=345: number analyzed (Participants) | 345
  Sitting Pulse Rate: Week 8, n=345 | 1.0 (9.98)
  Sitting Pulse Rate: Week 12, n=342: number analyzed (Participants) | 342
  Sitting Pulse Rate: Week 12, n=342 | 0.0 (9.52)
  Sitting Pulse Rate: Week 16, n=341: number analyzed (Participants) | 341
  Sitting Pulse Rate: Week 16, n=341 | -0.1 (10.08)
  Sitting Pulse Rate: Week 20, n=338: number analyzed (Participants) | 338
  Sitting Pulse Rate: Week 20, n=338 | -0.3 (9.44)
  Sitting Pulse Rate: Week 24, n=337: number analyzed (Participants) | 337
  Sitting Pulse Rate: Week 24, n=337 | -1.6 (9.83)
  Sitting Pulse Rate: Week 28, n=332: number analyzed (Participants) | 332
  Sitting Pulse Rate: Week 28, n=332 | -0.2 (9.58)
  Sitting Pulse Rate: Week 32, n=333: number analyzed (Participants) | 333
  Sitting Pulse Rate: Week 32, n=333 | -0.2 (9.74)
  Sitting Pulse Rate: Week 36, n=329: number analyzed (Participants) | 329
  Sitting Pulse Rate: Week 36, n=329 | -0.6 (9.60)
  Sitting Pulse Rate: Week 40, n=329: number analyzed (Participants) | 329
  Sitting Pulse Rate: Week 40, n=329 | -0.2 (9.56)
  Sitting Pulse Rate: Week 44, n=327: number analyzed (Participants) | 327
  Sitting Pulse Rate: Week 44, n=327 | -0.4 (9.80)
  Sitting Pulse Rate: Week 48, n=325: number analyzed (Participants) | 325
  Sitting Pulse Rate: Week 48, n=325 | -1.6 (9.65)
  Sitting Pulse Rate: Week 52, n=322: number analyzed (Participants) | 322
  Sitting Pulse Rate: Week 52, n=322 | 0.1 (9.56)
  Sitting Pulse Rate: Week 56, n=320: number analyzed (Participants) | 320
  Sitting Pulse Rate: Week 56, n=320 | -0.3 (9.79)
  Sitting Pulse Rate: Week 60, n=318: number analyzed (Participants) | 318
  Sitting Pulse Rate: Week 60, n=318 | -0.8 (9.54)
  Sitting Pulse Rate: Week 64, n=318: number analyzed (Participants) | 318
  Sitting Pulse Rate: Week 64, n=318 | -0.9 (9.63)
  Sitting Pulse Rate: Week 68, n=317: number analyzed (Participants) | 317
  Sitting Pulse Rate: Week 68, n=317 | -1.2 (9.51)
  Sitting Pulse Rate: Week 72, n=312: number analyzed (Participants) | 312
  Sitting Pulse Rate: Week 72, n=312 | -1.8 (10.07)
  Sitting Pulse Rate: Week 76, n=313: number analyzed (Participants) | 313
  Sitting Pulse Rate: Week 76, n=313 | -1.2 (9.65)
  Sitting Pulse Rate: Week 80, n=311: number analyzed (Participants) | 311
  Sitting Pulse Rate: Week 80, n=311 | -0.5 (10.08)
  Sitting Pulse Rate: Week 84, n=310: number analyzed (Participants) | 310
  Sitting Pulse Rate: Week 84, n=310 | -1.2 (9.80)
  Sitting Pulse Rate: Week 88, n=310: number analyzed (Participants) | 310
  Sitting Pulse Rate: Week 88, n=310 | -0.6 (10.12)
  Sitting Pulse Rate: Week 92, n=311: number analyzed (Participants) | 311
  Sitting Pulse Rate: Week 92, n=311 | -0.6 (9.36)
  Sitting Pulse Rate: Week 96, n=303: number analyzed (Participants) | 303
  Sitting Pulse Rate: Week 96, n=303 | -1.7 (10.61)
  Sitting Pulse Rate: Week 100, n=300: number analyzed (Participants) | 300
  Sitting Pulse Rate: Week 100, n=300 | -0.5 (9.81)
  Sitting Pulse Rate: Week 104, n=301: number analyzed (Participants) | 301
  Sitting Pulse Rate: Week 104, n=301 | -0.9 (10.45)
  Sitting Pulse Rate: Week 108, n=300: number analyzed (Participants) | 300
  Sitting Pulse Rate: Week 108, n=300 | -0.8 (10.04)
  Sitting Pulse Rate: Week 112, n=299: number analyzed (Participants) | 299
  Sitting Pulse Rate: Week 112, n=299 | -0.5 (9.60)
  Sitting Pulse Rate: Week 116, n=297: number analyzed (Participants) | 297
  Sitting Pulse Rate: Week 116, n=297 | -1.5 (9.33)
  Sitting Pulse Rate: Week 120, n=294: number analyzed (Participants) | 294
  Sitting Pulse Rate: Week 120, n=294 | -1.2 (10.27)
  Sitting Pulse Rate: Week 124, n=294: number analyzed (Participants) | 294
  Sitting Pulse Rate: Week 124, n=294 | -2.5 (10.27)
  Sitting Pulse Rate: Week 128, n=293: number analyzed (Participants) | 293
  Sitting Pulse Rate: Week 128, n=293 | -1.2 (10.00)
  Sitting Pulse Rate: Week 132, n=289: number analyzed (Participants) | 289
  Sitting Pulse Rate: Week 132, n=289 | -0.7 (9.20)
  Sitting Pulse Rate: Week 136, n=288: number analyzed (Participants) | 288
  Sitting Pulse Rate: Week 136, n=288 | -0.6 (10.55)
  Sitting Pulse Rate: Week 140, n=287: number analyzed (Participants) | 287
  Sitting Pulse Rate: Week 140, n=287 | -0.6 (9.71)
  Sitting Pulse Rate: Week 144, n=290: number analyzed (Participants) | 290
  Sitting Pulse Rate: Week 144, n=290 | -0.7 (9.72)
  Sitting Pulse Rate: Week 148, n=287: number analyzed (Participants) | 287
  Sitting Pulse Rate: Week 148, n=287 | -1.8 (9.82)
  Sitting Pulse Rate: Week 152, n=284: number analyzed (Participants) | 284
  Sitting Pulse Rate: Week 152, n=284 | -0.9 (10.45)
  Sitting Pulse Rate: Week 156, n=275: number analyzed (Participants) | 275
  Sitting Pulse Rate: Week 156, n=275 | -0.8 (9.83)
  Sitting Pulse Rate: Week 160, n=265: number analyzed (Participants) | 265
  Sitting Pulse Rate: Week 160, n=265 | -0.5 (10.42)
  Sitting Pulse Rate: Week 164, n=242: number analyzed (Participants) | 242
  Sitting Pulse Rate: Week 164, n=242 | -1.1 (11.07)
  Sitting Pulse Rate: Week 168, n=232: number analyzed (Participants) | 232
  Sitting Pulse Rate: Week 168, n=232 | -0.5 (11.25)
  Sitting Pulse Rate: Week 172, n=226: number analyzed (Participants) | 226
  Sitting Pulse Rate: Week 172, n=226 | -1.0 (9.80)
  Sitting Pulse Rate: Week 176, n=212: number analyzed (Participants) | 212
  Sitting Pulse Rate: Week 176, n=212 | -2.9 (9.57)
  Sitting Pulse Rate: Week 180, n=200: number analyzed (Participants) | 200
  Sitting Pulse Rate: Week 180, n=200 | -0.5 (10.01)
  Sitting Pulse Rate: Week 184, n=184: number analyzed (Participants) | 184
  Sitting Pulse Rate: Week 184, n=184 | -1.3 (9.89)
  Sitting Pulse Rate: Week 188, n=180: number analyzed (Participants) | 180
  Sitting Pulse Rate: Week 188, n=180 | -1.3 (10.38)
  Sitting Pulse Rate: Week 192, n=176: number analyzed (Participants) | 176
  Sitting Pulse Rate: Week 192, n=176 | -1.6 (10.37)
  Sitting Pulse Rate: Week 196, n=175: number analyzed (Participants) | 175
  Sitting Pulse Rate: Week 196, n=175 | -1.2 (9.79)
  Sitting Pulse Rate: Week 200, n=172: number analyzed (Participants) | 172
  Sitting Pulse Rate: Week 200, n=172 | -2.3 (11.03)
  Sitting Pulse Rate: Week 204, n=169: number analyzed (Participants) | 169
  Sitting Pulse Rate: Week 204, n=169 | -1.9 (10.67)
  Sitting Pulse Rate: Week 208, n=157: number analyzed (Participants) | 157
  Sitting Pulse Rate: Week 208, n=157 | -0.6 (10.64)
  Sitting Pulse Rate: Week 212, n=146: number analyzed (Participants) | 146
  Sitting Pulse Rate: Week 212, n=146 | -0.4 (10.09)
  Sitting Pulse Rate: Week 216, n=130: number analyzed (Participants) | 130
  Sitting Pulse Rate: Week 216, n=130 | -1.4 (10.49)
  Sitting Pulse Rate: Week 220, n=67: number analyzed (Participants) | 67
  Sitting Pulse Rate: Week 220, n=67 | -0.0 (11.13)
  Sitting Pulse Rate: Week 224, n=54: number analyzed (Participants) | 54
  Sitting Pulse Rate: Week 224, n=54 | -1.4 (13.19)
  Sitting Pulse Rate: Week 228, n=37: number analyzed (Participants) | 37
  Sitting Pulse Rate: Week 228, n=37 | -2.4 (10.57)
  Sitting Pulse Rate: Week 232, n=5: number analyzed (Participants) | 5
  Sitting Pulse Rate: Week 232, n=5 | -2.0 (16.63)
  Sitting Pulse Rate: Follow-up, n=306: number analyzed (Participants) | 306
  Sitting Pulse Rate: Follow-up, n=306 | -1.5 (10.72)

10. Secondary Outcome: Annualized Rate of On-treatment Exacerbations
Description: Exacerbations were defined as worsening of asthma which required use of systemic corticosteroids and/or hospitalization and/or Emergency Department visits. Data is presented as mean which is exacerbation rate/year. Exacerbation data are performed using a negative binomial model with covariates of region, annualized rate of exacerbations in the interval between MEA112997 and MEA115666 (as an ordinal variable) and baseline % predicted FEV1, and with logarithm of time on treatment as an offset variable.
Time Frame: Baseline (Week 0) to Week 240
Population: AT Population.
Measure: Mean (95% Confidence Interval); unit: Exacerbations per year
Arm/Group | Mepolizumab 100 mg
Number analyzed (Participants) | 347
Exacerbations per year | 0.68 [0.60 to 0.78]

11. Secondary Outcome: Mean Change From Baseline in Asthma Control Questionnaire (ACQ) Score
Description: The ACQ-5 is a five-item questionnaire, which was developed as a measure of participant' asthma control that was completed by the participant. The five questions enquire about the frequency and/or severity of symptoms (nocturnal awakening on waking in the morning, activity limitation, and shortness of breath, wheeze). The ACQ consists of 5 questions that are scored on a 7 point scale from 0 (totally controlled) to 6 (severely uncontrolled). The ACQ score was derived as mean of five questions: ACQ score = Question 1 (Q1)+Q2+Q3+Q4+Q5 divided by 5 where Q1, Q2,... Q5 are the scores of Q1, Q2, ..., Q5, respectively. The total score ranged from zero (no impairment/limitation) which indicated best condition to six (total impairment/ limitation) which indicated worst asthma. Baseline was Week 0. Change from Baseline was post-Baseline values minus Baseline values. Only those participants available at the specified time points were analyzed represented by n=X in the category titles.
Time Frame: Baseline (Week 0) to Week 240
Population: AT Population.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Mepolizumab 100 mg
Number analyzed (Participants) | 347
Scores on a Scale
  Week 12, n=341: number analyzed (Participants) | 341
  Week 12, n=341 | -0.47 (0.991)
  Week 24, n=335: number analyzed (Participants) | 335
  Week 24, n=335 | -0.55 (1.037)
  Week 36, n=327: number analyzed (Participants) | 327
  Week 36, n=327 | -0.56 (1.088)
  Week 48, n=324: number analyzed (Participants) | 324
  Week 48, n=324 | -0.55 (1.098)
  Week 60, n=317: number analyzed (Participants) | 317
  Week 60, n=317 | -0.58 (1.126)
  Week 72, n=311: number analyzed (Participants) | 311
  Week 72, n=311 | -0.51 (1.054)
  Week 84, n=308: number analyzed (Participants) | 308
  Week 84, n=308 | -0.54 (1.090)
  Week 96, n=301: number analyzed (Participants) | 301
  Week 96, n=301 | -0.44 (1.171)
  Week 112, n=297: number analyzed (Participants) | 297
  Week 112, n=297 | -0.51 (1.228)
  Week 124, n=293: number analyzed (Participants) | 293
  Week 124, n=293 | -0.66 (1.216)
  Week 136, n=287: number analyzed (Participants) | 287
  Week 136, n=287 | -0.58 (1.215)
  Week 148, n=286: number analyzed (Participants) | 286
  Week 148, n=286 | -0.54 (1.070)
  Week 164, n=240: number analyzed (Participants) | 240
  Week 164, n=240 | -0.59 (1.221)
  Week 176, n=211: number analyzed (Participants) | 211
  Week 176, n=211 | -0.49 (1.179)
  Week 188, n=178: number analyzed (Participants) | 178
  Week 188, n=178 | -0.40 (1.310)
  Week 200, n=171: number analyzed (Participants) | 171
  Week 200, n=171 | -0.45 (1.119)
  Week 216, n=130: number analyzed (Participants) | 130
  Week 216, n=130 | -0.42 (1.161)
  Week 228, n=37: number analyzed (Participants) | 37
  Week 228, n=37 | -0.47 (1.502)
  Follow-up, n=301: number analyzed (Participants) | 301
  Follow-up, n=301 | -0.53 (1.193)

12. Secondary Outcome: Mean Change From Baseline in Clinic Pre-bronchodilator Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 is forced expiratory volume in the first second. The volume of air that can be forced out in one second after taking a deep breath, an important measure of pulmonary function. Forced expiratory volume (FEV) measures how much air a person can exhale during a forced breath. FEV1 was measured by clinic spirometry. Baseline was Week 0. Change from Baseline was post-Baseline values minus Baseline values. Only those participants available at the specified time points were analyzed represented by n=X in the category titles.
Time Frame: Baseline (Week 0) to Week 240
Population: AT Population.
Measure: Mean (Standard Deviation); unit: Milliliters (mL)
Arm/Group | Mepolizumab 100 mg
Number analyzed (Participants) | 347
Milliliters (mL)
  Week 12, n=340: number analyzed (Participants) | 340
  Week 12, n=340 | 124 (346.9)
  Week 24, n=334: number analyzed (Participants) | 334
  Week 24, n=334 | 144 (335.0)
  Week 48, n=325: number analyzed (Participants) | 325
  Week 48, n=325 | 98 (395.2)
  Week 72, n=312: number analyzed (Participants) | 312
  Week 72, n=312 | 91 (405.5)
  Week 96, n=301: number analyzed (Participants) | 301
  Week 96, n=301 | 51 (385.8)
  Week 124, n=292: number analyzed (Participants) | 292
  Week 124, n=292 | 85 (395.5)
  Week 148, n=281: number analyzed (Participants) | 281
  Week 148, n=281 | 17 (370.2)
  Week 176, n=210: number analyzed (Participants) | 210
  Week 176, n=210 | 45 (352.2)
  Week 200, n=171: number analyzed (Participants) | 171
  Week 200, n=171 | 8 (375.7)
  Week 228, n=37: number analyzed (Participants) | 37
  Week 228, n=37 | -23 (331.9)

13. Secondary Outcome: Number of Participants With Positive Anti-mepolizumab Binding Antibodies (ADA) and Neutralizing Antibodies (NAb)
Description: Immunogenicity testing included two types of assays: a binding antibody assay (anti-drug antibody; ADA) and a neutralizing antibody (NAb) assay for participants who were tested positive in the ADA assay. Blood samples were collected for the determination of anti-mepolizumab antibodies, just prior to administration of mepolizumab. Samples that test positive for anti-mepolizumab antibodies were further tested for the presence of neutralizing antibody. Number of participants with positive highest value post-Baseline have been presented. Only those participants available at the specified time points were analyzed represented by n=X in the category titles.
Time Frame: Baseline (Week 0) to Week 240
Population: AT Population.
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 100 mg
Number analyzed (Participants) | 347
Participants
  Positive ADA result, n=346: number analyzed (Participants) | 346
  Positive ADA result, n=346 | 27
  Positive NAb result, n=27: number analyzed (Participants) | 27
  Positive NAb result, n=27 | 0

14. Secondary Outcome: Number of Participants Who Withdrew Due to Lack of Efficacy
Description: Lack of efficacy referred to failure of expected pharmacological action of Mepolizumab. Number of participants who withdrew due to lack of efficacy are presented.
Time Frame: Baseline (Week 0) to Week 240
Population: AT Population.
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 100 mg
Number analyzed (Participants) | 347
Participants | 11

15. Secondary Outcome: Number of Participants Requiring Hospitalizations Due to Adverse Events Including Asthma Exacerbations
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant or all events of possible drug induced liver injury with hyperbilirubinemia. Number of participants requiring hospitalization due to an on-treatment serious adverse event including asthma exacerbations are presented. On-treatment SAEs are the events occurring on/after the first dose of open-label mepolizumab date and before/on last dose of mepolizumab + 28 days.
Time Frame: Baseline (Week 0) to Week 240
Population: AT Population.
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 100 mg
Number analyzed (Participants) | 347
Participants | 71

16. Secondary Outcome: Number of Participants Who Withdrew Due to AE
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant or all events of possible drug induced liver injury with hyperbilirubinemia. Number of participants who withdrew due to AE are presented.
Time Frame: Baseline (Week 0) to Week 240
Population: AT Population.
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 100 mg
Number analyzed (Participants) | 347
Participants | 19

ADVERSE EVENTS:
Time Frame: The on-treatment AEs and on-treatment SAEs are the events which happened on/after the first dose of open label mepolizumab date and before/on last dose of mepolizumab date + 28 days (up to 240 weeks)
Description: AE and SAE were collected for all participants within the As Treated Population which comprised of all participants who received at least one dose of open label mepolizumab.
Arm/Group | Mepolizumab
All-Cause Mortality (participants affected / at risk) | 6/347
Serious Adverse Events (participants affected / at risk) | 79/347
Other Adverse Events (participants affected / at risk) | 314/347
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mepolizumab (N=347)
Asthma (Respiratory, thoracic and mediastinal disorders) | 33
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 6
Cellulitis (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 2
Abscess limb (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Myelitis (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Chronic gastritis (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Gastric polyps (Gastrointestinal disorders) | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Atrial tachycardia (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Epilepsy (Nervous system disorders) | 2
Sciatica (Nervous system disorders) | 2
Cerebral haemorrhage (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Peroneal nerve palsy (Nervous system disorders) | 1
Spinal claudication (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chills (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Sudden death (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Cholestasis (Hepatobiliary disorders) | 1
Hepatocellular injury (Hepatobiliary disorders) | 1
Hypertension (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Anaphylactic shock (Immune system disorders) | 1
Blood glucose increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Bladder prolapse (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Cervical polyp (Reproductive system and breast disorders) | 1
Rectocele (Reproductive system and breast disorders) | 1
Lymphocytosis (Blood and lymphatic system disorders) | 1
Basedow's disease (Endocrine disorders) | 1
Thyroid mass (Endocrine disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mepolizumab (N=347)
Viral upper respiratory tract infection (Infections and infestations) | 169
Upper respiratory tract infection (Infections and infestations) | 81
Bronchitis (Infections and infestations) | 73
Sinusitis (Infections and infestations) | 57
Influenza (Infections and infestations) | 43
Respiratory tract infection (Infections and infestations) | 38
Lower respiratory tract infection (Infections and infestations) | 31
Gastroenteritis (Infections and infestations) | 27
Pharyngitis (Infections and infestations) | 24
Urinary tract infection (Infections and infestations) | 24
Rhinitis (Infections and infestations) | 23
Respiratory tract infection viral (Infections and infestations) | 20
Viral infection (Infections and infestations) | 18
Ear infection (Infections and infestations) | 15
Acute sinusitis (Infections and infestations) | 14
Cystitis (Infections and infestations) | 13
Nasopharyngitis (Infections and infestations) | 13
Oral candidiasis (Infections and infestations) | 13
Asthma (Respiratory, thoracic and mediastinal disorders) | 69
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 36
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 22
Productive cough (Respiratory, thoracic and mediastinal disorders) | 12
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Back pain (Musculoskeletal and connective tissue disorders) | 63
Arthralgia (Musculoskeletal and connective tissue disorders) | 58
Pain in extremity (Musculoskeletal and connective tissue disorders) | 40
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 18
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14
Headache (Nervous system disorders) | 99
Dizziness (Nervous system disorders) | 23
Sciatica (Nervous system disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 26
Toothache (Gastrointestinal disorders) | 22
Abdominal pain (Gastrointestinal disorders) | 17
Nausea (Gastrointestinal disorders) | 17
Abdominal pain upper (Gastrointestinal disorders) | 15
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 14
Dyspepsia (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 11
Injection site reaction (General disorders) | 42
Fatigue (General disorders) | 12
Laceration (Injury, poisoning and procedural complications) | 15
Contusion (Injury, poisoning and procedural complications) | 13
Ligament sprain (Injury, poisoning and procedural complications) | 11
Hypertension (Vascular disorders) | 32
Cataract (Eye disorders) | 14
Hypersensitivity (Immune system disorders) | 13
Rash (Skin and subcutaneous tissue disorders) | 12
Hypercholesterolaemia (Metabolism and nutrition disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-06-19): https://cdn.clinicaltrials.gov/large-docs/59/NCT01691859/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-06): https://cdn.clinicaltrials.gov/large-docs/59/NCT01691859/SAP_001.pdf